CLINICAL TRIAL: NCT00449514
Title: Prospective Randomized Study of Ovulation Induction Using Either Tamoxifen or Clomiphene Citrate for Women Who Had Thin Endometrium During Previous Treatment With Clomiphene Citrate
Brief Title: Tamoxifen Compared With Clomiphene Citrate for Women Who Had Thin Endometrium Women Under Clomiphene in a Previous Cycle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: tamoxi vs clomiphene.CTIL
Record Dates: First submitted 2007-03-18; First posted 2007-03-20 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-05

CONDITIONS: Infertility
Keywords: infertility; ovulation dysfunction; endometrium; tamoxifen; clomiphene citrate
MeSH Terms: conditions — Infertility | interventions — Tamoxifen; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: tamoxifen
Drug: clomiphene citrate

SUMMARY:
About 10-15% of all couples attempting to conceive will not become pregnant within one year. Among those, the majority will have ovulatory dysfunction, mild male infertility or unexplained infertility. The traditional first line therapy for those couples is ovulation induction or superovulation using clomiphene citrate. Probably due to anti-estrogenic effects of this agent will, some patients will have a thin endometrium as measured by sonography at the time of ovulation. This phenomenon may be associated with a lower chance to conceive. Tamoxifen is a similar molecule that has been used to clomiphene citrate that has been shown to be equally effective to clomiphene in ovulation induction. Preliminary observations showed that tamoxifen does not cause a negative effect on the endometrium as compared with clomiphene, and may increase the chance to conceive in those patients who have a thin endometrium under clomiphene.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary infertility due to:
* Ovulatory dysfunction
* Mild male infertility
* Unexplained infertility
* Endometrium < 6 mm at time of hCG during previous treatment with clomiphene citrate
* Age 18-35

Exclusion Criteria:

* Serious adverse effects under clomiphene citrate or known sensitivity to either tamoxifen or clomiphene citrate

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-05

PRIMARY OUTCOMES:
Pregnancy rate
delivery rate

SECONDARY OUTCOMES:
endometrium thickness
percentage of ovulation
number of follicles

CONTACTS AND LOCATIONS:
Overall Officials: Avi Tsafrir, MD, Principal Investigator — Department of Obstetrics and Gynecology, Shaare-Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Shaare-Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Steiner AZ, Terplan M, Paulson RJ. Comparison of tamoxifen and clomiphene citrate for ovulation induction: a meta-analysis. Hum Reprod. 2005 Jun;20(6):1511-5. doi: 10.1093/humrep/deh840. Epub 2005 Apr 21. PMID 15845599